CLINICAL TRIAL: NCT05801822
Title: Prevalence of Sub-clinical Hypothyroidism Among Pregnant Women During First Trimester: Cross Sectional Study.
Brief Title: Screening of Subclinical Hypothyroidism in Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amira Mostafa Mahmoud, resident doctor, Sohag University
Other Study IDs: Soh-Med-23-03-02MS
Record Dates: First submitted 2023-03-25; First posted 2023-04-06 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Subclinical Hypothyroidism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum T.S.H level test — , the blood samples will be collected and to be assessed for the routine antenatal screening CBC, random blood sugar, HBV and HIV, the same blood sample will be used to asses TSH level.

SUMMARY:
this study may help the physicians to evaluate the practice of universal screening of sub-clinical hypothyroidism and thyroid-stimulating hormone level. Detection of sub-clinical hypothyroidism early in pregnancy through thyroid-stimulating hormone sampling in the first trimester will allow achieving proper management and better maternal and neonatal outcome of these patients.

DETAILED DESCRIPTION:
This is a cross-sectional study will be carried out on women attending Obstetrics Outpatient Clinic in Sohag University Hospitals between April and 1st December 2023 for the booking antenatal care visit and to be invited to enroll in the study. The attending physician will explain the nature of the study to the cases, the blood samples will be collected and to be assessed for the routine antenatal screening complete blood count, random blood sugar, hepatitis B virus and HIV, the same blood sample will be used to asses TSH level.

ELIGIBILITY:
Inclusion Criteria:

* Age group 18 years to 45 years.
* first trimester pregnant women.

Exclusion Criteria:

* Women with known thyroid disorders or previous thyroidectomy.
* Pregnant women with hyperemesis gravidarum.
* Molar pregnancy.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — subclinical hypothyroidism in pregnant women
Study Population: This is a cross-sectional study will be carried out on women attending Obstetrics Outpatient Clinic in Sohag University Hospitals for the booking antenatal care visit.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
diagnosis of subclinical hypothyroidism early in pregnancy | in the first trimester of pregnancy ( first 12 weeks)
  by serum TSH level

CONTACTS AND LOCATIONS:
Overall Officials: Amira M Mahmoud, bachelor, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: Undecided